CLINICAL TRIAL: NCT02174003
Title: Whole Body Hyperthermia Registry Study
Status: Terminated | Type: Observational
Why Stopped: Investigator transferred to the University of Wisconsin - Madison
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Other Study IDs: 1406365027
Record Dates: First submitted 2014-06-23; First posted 2014-06-25 (Estimated); Last update posted 2025-07-31 (Actual); Status verified 2015-07

CONDITIONS: Depression; Anxiety; PTSD; Fibromyalgia; Chronic Fatigue Syndrome
Keywords: whole body hyperthermia; depression; fibromyalgia; rheumatoid arthritis; perimenopausal symptoms; open treatment
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic; Fibromyalgia; Fatigue Syndrome, Chronic; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Open Treatment Group: The Open Treatment Group (all participants in this study) will receive the active / WBH treatment in an open fashion.
  Interventions: Device: High intensity whole-body infrared heating

INTERVENTIONS:
Device: High intensity whole-body infrared heating — The Whole Body Hyperthermia system uses water-filtered infrared-A (wIRA) heat radiation. The rise in the body's core temperature is correspondingly rapid and well-tolerated. There are two phases of the thermal challenge, 1) Irradiation phase during which the patient lies recumbent with his/her head positioned outside the tent. The wIRA irradiators are arranged above the exposed upper part of the body; and 2) Heat retention phase during which the patient lies in the chamber with the walls of the tent positioned to retain heat. Core body temperatures will be raised to those comparable to a mild fever 37.8-38.5°C.
  Other Names: WBH

SUMMARY:
This protocol will allow for the implementation of a research registry pertaining to Whole Body Hyperthermia (WBH) use in various subject populations. The primary objective of the proposed study is to determine if WBH can have beneficial effects in various subject populations currently experiencing numerous other comorbidities, and the duration of the effect(s).

This protocol is intended to become a secondary resort for individual's interested in receiving a Hyperthermia treatment for potential beneficial gain related to symptoms stemming from comorbidities other than depression (i.e. Fibromyalgia, Perimenopausal symptoms, arthritis, etc). Due to the fact that no external research funding has been acquired for this broad application this protocol is intended to charge a fee for cost covering purposes only.

The registry trial will not be limited to only include individuals with major depressive disorder, however, this protocol will allow for an expanded use in all populations (while still excluding subjects based on safety parameters). We will monitor subject's physiological and clinical outcomes (if applicable) from a single Whole Body Hyperthermia treatment in an open fashion (no placebo/control condition). This registry study will include safety assessments 5 days prior to WBH, the day of WBH and 1 week following WBH.

DETAILED DESCRIPTION:
The WBH procedure proposed in this protocol has been rigorously researched in subjects with Major Depressive Disorder (MDD), and there are little to no preliminary data pertaining to WBH use in populations outside of depression studies. In preliminary studies in Europe and a rigorously tested clinical trial being conducted at the University of Arizona (NCT01625546), a single exposure to WBH resulted in a decrease in depressive symptoms as measured using the German version of the CES-D depression scale 5 days later (in the study in Switzerland) and using the HamD rating scale 7 days later in the UA study. All research applications thus far have resulted in minimal adverse effects to study subjects.

During the conduct of research protocol 12-0147-04/NCT01625546 (WBH in subjects with Major Depression) our research site has been contacted by numerous individuals across the country asking if they can participate in our clinical trial. However due to the rigorous inclusion/exclusion criteria necessary for data collection, these individuals cannot be offered the research treatment. This protocol is intended to become a secondary resort for these individual's interested in receiving a Hyperthermia treatment for potential beneficial gain related to symptoms stemming from other comorbidities (i.e. Fibromyalgia, Perimenopausal symptoms, arthritis, etc). In fact, over the course of this study, several individuals who suffer from fibromyalgia, rheumatoid arthritis and other similar afflictions have, in discussions with study staff at screening, indicated that they have previously researched infrared heating and whole body hyperthermia and found that it was helpful to many people with these afflictions. As such, they are interested in being a part of the study in order to receive treatment that might help ease their pain from these afflictions in addition to the depression symptoms they are experiencing, given that depression is often a co-morbidity of these illnesses. Due to the fact that no external research funding has been acquired for this broad application, this protocol intended to charge a fee for cost covering purposes only.

The registry trial will not be limited to only include individuals with MDD, however this protocol will allow for an expanded use in all populations (while still excluding subjects based on safety parameters). We will monitor subject's physiological and clinical outcomes (if applicable) from a single Whole Body Hyperthermia treatment in an open fashion (no placebo/control condition). This registry study will include safety assessments 5 days prior to WBH, the day of WBH and 1 week following WBH.

Costs for Participating in the Study:

The WBH session is an investigational procedure, one approved for limited testing by the Food and Drug Administration (FDA) but not in general use. In addition to your time, you will be charged a fee of $800 for cost covering purposes only. The cost for this open treatment hyperthermia session will cover departmental staff time, clinical space, research materials, and overhead fees. You may pay with cash, check, or credit card. If you wish to pay with a credit card, a 3% fee will be assessed to cover credit card processing fees. All payments will be made to the Department of Psychiatry and will be processed by our Departmental business office.

The payment may be broken into 2 tiers:

Screening: $200 WBH Procedure: $600 If you qualify for WBH procedure the remaining $600 will be due prior to completion of the procedure.

If you pay in full and it is determined you do not qualify for the study, you will be reimbursed less any amount needed to cover procedures performed (i.e. screening).

Future WBH Treatment Sessions:

If you wish to undergo another WBH procedure, you may do so without have to repeat screening bloods and EKG's within 1 year of the original screen, so long as you report no significant changes in your health history to the study staff. You will not be charged for screening procedures for subsequent WBH procedures. Those individuals who have participated in previous WBH protocols will be considered eligible without need for a re-screen within 1 year of their original screening procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients aged 18+.
* Able to understand the nature of the study and able to provide written informed consent prior to conduct of any study procedures.
* Able to communicate in English or Spanish with study personnel.

Exclusion Criteria:

* If patient has a medical condition or disorder that:

  * Is unstable and clinically significant, or:
  * Could, in the investigator's opinion, interfere with the accurate assessment of safety or efficacy of the procedure, including:
* Individuals who are using prescription drugs that may impair thermoregulatory cooling,
* Individuals with cardiovascular conditions or problems (uncontrolled hypertension, congestive heart failure, or documented evidence of coronary artery disease)
* Individuals with chronic conditions/diseases associated with a reduced ability initiate thermoregulatory cooling, including Parkinson's, multiple sclerosis, central nervous system tumors, and diabetes with neuropathy,
* Individuals with a fever the day of study intervention (if so, they will be rescheduled),
* Individuals with hypersensitivity to heat,
* Individuals with enclosed infections, be they dental, in joints, or in any other tissues,
* Women who are pregnant Obesity and overall size of subject.
* It will be up to the PI's discretion will consider BMI, waist circumference, and body fat composition when determining eligibility and safety of the individual.
* History of peripheral circulatory disease, for example peripheral vascular disease, deep vein thrombosis (DVT), or lymphedema.
* History of stroke, epilepsy or cerebral aneurisms
* Diabetes mellitus types I or II.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For the purposes of this study we will enroll subjects 18 years and older to undergo a Hyperthermia session in an open fashion. We expect approximately 20-30 subjects per year to undergo this open hyperthermia treatment. Subjects must be medically healthy enough to be able to undergo the Hyperthermia session, all exclusion criteria listed below address what is deemed "medically healthy".
  Inclusion into this study will require that the minimum safety standards described in the eligibility criteria, there will be no inclusion of children, pregnant women, mentally impaired individuals, or prisoners in this registry. Subjects who appear to have Major Depressive Disorder will be referred to Protocol 12-0147-01 due to the specific aims pertaining directly to depressive symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2014-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in depression scores over time [Inventory of Depressive Symptomatology-Self Report (IDS-SR)] | Screening, WBH treatment day and 1 week following treatment.
  Percent change in scores between baseline and subsequent assessments will be assessed

SECONDARY OUTCOMES:
Change in Positive and Negative Affect | Screening, WBH treatment and 1 week following WBH treatment
  Percent change in positive and negative affect will be assessed between baseline and subsequent assessments using the Positive and Negative Affect Schedule (PANAS)
Change in Morning / Evening Questionnaire | Screening, WBH Treatment day, 1 week following WBH Treatment
  Percent change in morning versus evening behavioral preferences will be assessed between baseline and subsequent assessments using the Morningness and Eveningness Questionnaire (MEQ).
Change in Quality of Life | Screening, WBH Treatment Day and 1 week following WBH treatment
  Percent change in scores using the Quality of Life Enjoyment and Satisfaction (Q-LESQ-SF) questionnaire.
Change in functional impairment | Screening, WBH Treatment Day and 1 week following WBH treatment day
  Percent change in score on the Sheehan Disability Scale to assess improvements in work/school, social and family life.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Raison, MD, Principal Investigator — University of Arizona, Department of Psychiatry, College of Medicine
Locations (1):
- University of Arizona, Tucson, Arizona, United States